CLINICAL TRIAL: NCT04024683
Title: The Effect of the Ultrasound-guided Serratus Anterior Plane Block in Combinaison With Thoracic Paravertebral cathéter Versus Thoracic Paravertebral Cather for Perioperative Analgesia in Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Bouhemad - BEAL 2019
Record Dates: First submitted 2019-07-15; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Thoracic Surgery
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Serratus block group: Realization of a serratus block and para-vertebral catheter
  Interventions: Procedure: Serratus block with ropivacaine 2mg/ml
- Control group: Realization of a para-vertebral catheter

INTERVENTIONS:
Procedure: Serratus block with ropivacaine 2mg/ml — The serratus block was made using a 50 mm needle with ultrasound guidance. It was performed supine, the ultrasound probe identifying the 3, 4 or 5th intercostal space and then the needle was introduced under ultrasound control
  Groups: Serratus block group

SUMMARY:
Introduction

The paravertebral catheter has been shown to be effective in controlling postoperative pain, but has never been associated with the deep dentate block in thoracic surgery. The objective of this study was to compare the efficacy of single-dose deep dentate block-level postoperative pain control in combination with a continuous perfusion paravertebral catheter versus continuous perfusion paravertebral catheter alone in controlled thoracic surgery.

Materials and methods

We retrospectively included 159 ASA I-III major patients who underwent scheduled thoracic surgery in the operating theater of Dijon University Hospital, between March and November 2018. All patients benefited from the same anesthetic protocol routinely used in controlled thoracic surgery. They were included in two groups: deep serrate deep group (GS) with a deep serrated deep serrate block immediately after orotracheal intubation with 0.2% Ropivacaine at 0.75 mg / kg and paravertebral catheter placed by the surgeon and put in charge at the fall of the surgical drapes versus control group (GC) benefiting from a paravertebral catheter alone. The primary endpoint was 24-hour morphine equivalent consumption. The criteria for secondary judgments were intraoperative remifentanil consumption, VAS at 0h, 24h and 48h, morphine consumption at 0h, 48h and the profile of the various complications. The morphine equivalent was calculated according to an equivalence table with reference to Oxycodone per os. Quantitative data are presented in median and standard deviation and were compared by Student's t-test or Wilcoxon test.

ELIGIBILITY:
Inclusion Criteria:

* We included all patients over the age of 18 who met the classification criteria of the American Society of Anesthesiology (ASA) and had thoracic surgery in the operating theater of Dijon University Hospital

Exclusion Criteria:

* Exclusion criteria were ASA 4 or higher, pregnant or breastfeeding women, minor patients, patients not able to use morphine PCA, and patients with chronic algia.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with thoracic surgery in the operating theater of Dijon University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
consumption of morphine equivalence | 24 hours

SECONDARY OUTCOMES:
intraoperative remifentanil consumption, | 48 hours
visual analogue scale | 48 hours
morphine consumption | 48 hours
intraoperative complications | Day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France